CLINICAL TRIAL: NCT05239013
Title: Safety and Tolerability of Topical Nitroglycerin to Dilate the Radial Artery Prior to Transradial Coronary Angiography
Brief Title: Safety and Tolerability of Nitro for Radial Artery Dilation
Acronym: RADial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RADial
Record Dates: First submitted 2022-02-07; First posted 2022-02-14 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Artery; Dilatation
Keywords: cardiac catheterization; transradial approach; nitroglycerin
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Subjects who receive the intervention
  Interventions: Drug: Nitroglycerin ointment

INTERVENTIONS:
Drug: Nitroglycerin ointment — 2 cm (30mg) of 2% nitroglycerin applied 2 cm from the styloid process of the anterior forearm
  Other Names: Nitropaste

SUMMARY:
Phase 1, single-center, open-label clinical study to assess the safety and efficacy of topical nitroglycerin on dilation of the radial artery. Subjects will receive nitroglycerin ointment prior to scheduled PCI and radial artery measurements will be performed to determine mean increase in radial artery diameter at several time points. There will be 20 subjects enrolled in this study.

DETAILED DESCRIPTION:
This is a phase I study evaluating the safety, tolerability, and efficacy of topical nitroglycerin prior to percutaneous coronary intervention (PCI). Although the ultimate plan is to evaluate this intervention vs placebo, it is important to first determine whether topical nitroglycerin not only is safe for patients, but whether it effectively dilates the radial artery. Given that patients who receive topical nitroglycerin applied to the chest for other reasons (angina or acute coronary syndrome, hypertension, etc) have reported headaches and/or have experienced decreased blood pressure, it is important to determine whether these noted side effects are present when nitroglycerin ointment is applied to the arm. Prior to initiating any study procedures, we will perform a Barbeau test to determine normal blood flow through the radial artery and collateral circulation from the ulnar artery through the palmar arch. After the ointment is applied, we will also be measuring the dimensions of the radial artery for the degree of dilation in order to determine whether topical nitroglycerin is indeed a possible method for increasing the rate of PCI performed using the transradial approach (TRA).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo PCI using TRA in the cardiac catheterization laboratory

Exclusion Criteria:

1. Known nitrate allergy
2. Baseline hypotension with systolic blood pressure <90mmHg
3. Absence of radial artery blood flow in one or both arms
4. Presence or history of liver, rheumatologic, or chronic kidney disease
5. Current treatment with any vasodilator therapy (eg. Sildenafil)
6. Radial artery catheterization <30 days prior to enrollment
7. Active site infection
8. AV-fistula or prior radial artery harvest for bypass surgery
9. Abnormal Barbeau test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 45 minutes
  Changes in blood pressure measured by upper arm cuff pressure
Incidence of headache | 45 minutes
  Rate and severity of headache, determined by subject-reported symptoms.
Hematoma | 45 minutes
  Incidence of forearm hematoma development

SECONDARY OUTCOMES:
Radial artery dilation | 45 minutes
  Change in radial artery dilation, measured by radial artery diameter using high-frequency (13MHz) linear array transducer 2cm proximal to the radial styloid process at 15 and 30 minute time points.
Punctures required | 45 minutes
  Number of radial artery punctures/attempts
Transradial conversions to transfemoral approach | 45 minutes
  Number of conversions to transfemoral approach

CONTACTS AND LOCATIONS:
Overall Officials: David Fischman, M.D., Principal Investigator — Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Background] Beyer AT, Ng R, Singh A, Zimmet J, Shunk K, Yeghiazarians Y, Ports TA, Boyle AJ. Topical nitroglycerin and lidocaine to dilate the radial artery prior to transradial cardiac catheterization: a randomized, placebo-controlled, double-blind clinical trial: the PRE-DILATE Study. Int J Cardiol. 2013 Oct 3;168(3):2575-8. doi: 10.1016/j.ijcard.2013.03.048. Epub 2013 Apr 10. PMID 23582415
- [Background] Caputo RP, Tremmel JA, Rao S, Gilchrist IC, Pyne C, Pancholy S, Frasier D, Gulati R, Skelding K, Bertrand O, Patel T. Transradial arterial access for coronary and peripheral procedures: executive summary by the Transradial Committee of the SCAI. Catheter Cardiovasc Interv. 2011 Nov 15;78(6):823-39. doi: 10.1002/ccd.23052. Epub 2011 May 4. PMID 21544927
- [Background] Divakaran S, Loscalzo J. The Role of Nitroglycerin and Other Nitrogen Oxides in Cardiovascular Therapeutics. J Am Coll Cardiol. 2017 Nov 7;70(19):2393-2410. doi: 10.1016/j.jacc.2017.09.1064. PMID 29096811
- [Background] Jolly SS, Amlani S, Hamon M, Yusuf S, Mehta SR. Radial versus femoral access for coronary angiography or intervention and the impact on major bleeding and ischemic events: a systematic review and meta-analysis of randomized trials. Am Heart J. 2009 Jan;157(1):132-40. doi: 10.1016/j.ahj.2008.08.023. Epub 2008 Nov 1. PMID 19081409
- [Background] Majure DT, Hallaux M, Yeghiazarians Y, Boyle AJ. Topical nitroglycerin and lidocaine locally vasodilate the radial artery without affecting systemic blood pressure: a dose-finding phase I study. J Crit Care. 2012 Oct;27(5):532.e9-13. doi: 10.1016/j.jcrc.2012.04.019. Epub 2012 Jun 12. PMID 22699036
- [Background] Manoukian SV, Feit F, Mehran R, Voeltz MD, Ebrahimi R, Hamon M, Dangas GD, Lincoff AM, White HD, Moses JW, King SB 3rd, Ohman EM, Stone GW. Impact of major bleeding on 30-day mortality and clinical outcomes in patients with acute coronary syndromes: an analysis from the ACUITY Trial. J Am Coll Cardiol. 2007 Mar 27;49(12):1362-8. doi: 10.1016/j.jacc.2007.02.027. Epub 2007 Mar 9. PMID 17394970
- [Background] Riegel B, Heywood G, Jackson W, Kennedy A. Effect of nitroglycerin ointment placement on the severity of headache and flushing in patients with cardiac disease. Heart Lung. 1988 Jul;17(4):426-31. PMID 3134314
- [Background] Wester RC, Noonan PK, Smeach S, Kosobud L. Pharmacokinetics and bioavailability of intravenous and topical nitroglycerin in the rhesus monkey: estimate of percutaneous first-pass metabolism. J Pharm Sci. 1983 Jul;72(7):745-8. doi: 10.1002/jps.2600720708. PMID 6411893